CLINICAL TRIAL: NCT03686839
Title: Importance of Exploring Feasibility and Acceptability in Application of EEG Neurofeedback in Older Adults With Mild Cognitive Impairment
Brief Title: Feasibility Study of Neurofeedback Training for Older Adults With Mild Cognitive Impairment
Acronym: Neurofeedel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabienne Marlats (Other)
Responsible Party: Sponsor-Investigator, Fabienne Marlats, Neuropsychologist, Broca Hospital
Organization: Broca Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LUS2EEGNF
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Mild Cognitive Impairment, So Stated
Keywords: Neurofeedback; Acceptance technology; Electroencephalography; MCI
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: no randomized, no controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMR neurofeedback training to MCI (Experimental): Sensorimotor rhythm neurofeedback protocol consisted of 20 individual sessions, twice a week, during 11 weeks maximum. For each subject MCI, NF was planned and conducted by a neuropsychologist experienced in neurophysiology and neurofeedback. Each session lasted 1h10-15min and was conducted as follows:
  1. Preparation and installation of the electrodes, verification of the impedance, adjustment of the calibration and thresholds (15 minutes).
  2. NF training (tasks and video described below) (45 minutes).
  3. Feedback and debriefing about the session (15 minutes).
  Interventions: Behavioral: SMR neurofeedback training to MCI

INTERVENTIONS:
Behavioral: SMR neurofeedback training to MCI — SMR neurofeedback training consisted to increase the synaptic strengths and sensitivity within this network. Electroencephalography signals for SMR/theta ratio training was recorded at channel Cz according to the International 10-20 system. Theta rhythm was also recorded and, in this case, SMR was stimulated while theta waves were suppressed. A 32 channels system (EEGDigitrack Biofeedback plus module, Inc Elmiko Medical) was used for SMR/theta neurofeedback training.
  Other Names: SMR

SUMMARY:
This is a non-pharmacological study evaluating the feasibility of a neurofeedback training program in elderly with mild cognitive impairment (MCI) according to recruitment, retention, attendance, acceptability data.

DETAILED DESCRIPTION:
Neurofeedback (NF) can be counted amongst promising techniques to improve cognitive functioning if the principles of application are seriously respected, whilst recognizing the necessary adaptation to the conditions of patients with Mild Cognitive Impairment (MCI). This study examined the feasibility and acceptability of an electroencephalography neurofeedback training protocol in a sample group of older adults with MCI in order to identify the necessary conditions for an improved neurofeedback application. Participants performed an electroencephalography recording, a battery of neuropsychological tests before the neurofeedback training program (T0), following the neurofeedback training program (T2) and 1-month follow-up (T3). A questionnaire about motivation, opinions of technical aspects of NF and feeling of cognitive improvement was administered at T0 and T2.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild Cognitive Impairment
* Absence of history of alcohol or other substance consumption

Exclusion Criteria:

* Psychiatric and neurological disorders
* sensory and/or motor deficit.
* involving in another cognitive intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Neurofeedback Technology Acceptation Questionnaire | Assessment was at 2 months immediately after the Neurofeedback intervention
  Neurofeedback Technology Acceptation Questionnaire assessed the participants' opinions face to the electroencephalography neurofeedback intervention with 33 questions. The mode of administration was a personal interview with the investigator, the type of questions was closed-ended (for binary variable yes or no). Answers were analyzed with the Multiple Correspondence Analysis to visualize associations and similarities among participants and answers to Questionnaire. An unsupervised hierarchical clustering was performed using the Euclidean distance and Ward's method. Clusters were defined graphically using dendrogram.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie AR Rigaud, Professor, Study Director — Broca University Hospital
Locations (1):
- Anne-Sophie Rigaud, Paris, France

IPD SHARING:
Plan to Share IPD: No